CLINICAL TRIAL: NCT00842361
Title: A 6-week, Randomised, Multi-centre, Open-labelled, Parallel Group, Exploratory Trial to Investigate the Safety of SIAC Compared to Mix30 (NovoRapid®30Mix) on a Twice Daily Regimen in Subjects With Type 2 Diabetes Mellitus
Brief Title: Comparison of NN5401 Versus Biphasic Insulin Aspart 30 on a Twice Daily Regimen in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3570; JapicCTI-090712 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mix30 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30
- SIAC (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — The insulin NN5401 (insulin degludec/insulin aspart) injected subcutaneously immediately before breakfast and dinner.
  Arms: SIAC
Drug: biphasic insulin aspart 30 — The insulin (biphasic insulin aspart 30) injected subcutaneously immediately before breakfast and dinner.
  Arms: Mix30

SUMMARY:
This trial is conducted in Japan. The aim of this clinical trial is to investigate the safety (with emphasis on hypoglycaemia) after switching from long-acting insulin analogue/intermediate-acting insulin or pre-mixed insulin/pre-mixed insulin analogue on a twice daily regimen to NN5401 (SIAC, insulin degludec/insulin aspart) on a twice daily regimen in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus
* Current treatment using a long-acting insulin analogue/intermediate-acting insulin preparation (except insulin glargine) or a pre-mixed insulin/insulin analogue preparation (except Mix30) on a twice daily regimen for at least 12 weeks, with stable insulin dose for the last 4 weeks (a brand of insulin preparation and dosing regimen has not been changed in the preceding 12 weeks)
* HbA1c below 10.0%
* Body Mass Index (BMI) < 30.0 kg/m^2

Exclusion Criteria:

* Known hypoglycaemia unawareness or recurrent major hypoglycaemia
* Current treatment with total insulin dose of more than 100 U or IU/day
* Current treatment or expected to start treatment with systemic corticosteroid
* Treatment with oral anti-diabetic drugs (OADs: including alpha-glucosidase inhibitor and insulin sensitizer [thiazolidinedione: TZD]) within the last 12 weeks prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk Pharma Ltd.
Locations (8):
- Japan (8):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Sendai
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tagajō-shi

REFERENCES:
- [Result] Onishi Y, Yamada K, Zacho J, Ekelund J, Iwamoto Y. Insulin degludec/insulin aspart vs biphasic insulin aspart 30 twice daily in Japanese patients with type 2 diabetes: A randomized controlled trial. J Diabetes Investig. 2017 Mar;8(2):210-217. doi: 10.1111/jdi.12569. Epub 2016 Oct 7. PMID 27560769
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 sites in Japan
Groups:
- SIAC: Soluble insulin basal analogue combination (SIAC, 70 volume percent insulin degludec, 600 nmol/ml and 30 volume percent insulin aspart [IAsp], 600 nmol/ml) was given subcutaneously twice daily immediately before breakfast and dinner for 6 weeks. Insulin doses were individually adjusted
- Mix30: Biphasic insulin aspart (IAsp) 30 (Mix30) (i.e., 30% IAsp and 70% protamine-crystallised IAsp) was given subcutaneously twice daily immediately before breakfast and dinner for 6 weeks. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | SIAC | Mix30
Started | 33 | 33
Exposed | 33 | 32 (One subject withdrew prior to exposure to trial drug)
Completed | 32 | 31
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Unclassified | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIAC | Mix30 | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.4) | 64.7 (11.2) | 64.5 (9.8)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 24 | 18 | 42
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.36 (0.86) | 7.44 (0.84) | 7.40 (0.84)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/L] | 144.6 (36.4) | 140.8 (38.6) | 142.7 (37.3)
Body weight [Mean (Standard Deviation); unit: kg] | 61.22 (9.88) | 57.32 (7.94) | 59.30 (9.12)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major and Minor Hypoglycaemic Episodes
Description: Rate of major and minor hypoglycaemic episodes per patient year (1year=365.25days) of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose ≤ 55 mg/dL.
Time Frame: Week 0 to Week 6 + 5 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes /year of patient exposure
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
Episodes /year of patient exposure
  Major | 0 | 0
  Minor | 13.63 | 21.83

2. Primary Outcome: Rate of Nocturnal Major and Minor Hypoglycaemic Episodes
Description: Rate of nocturnal major and minor hypoglycaemic episodes per patient year (1year=365.25days) of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose ≤ 55 mg/dL. Episodes were defined as nocturnal if the time of onset was between 23:00 and 05:59 (both inclusive).
Time Frame: Week 0 to Week 6 + 5 days follow up
Population: as for outcome 1
Measure: Number; unit: Episodes /year of patient exposure
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
Episodes /year of patient exposure
  Major | 0 | 0
  Minor | 0.99 | 2.03

3. Secondary Outcome: Number of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to number of adverse events. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 6 + 5 days follow up
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
events
  Adverse events (AEs) | 13 | 8
  Serious AEs | 1 | 0
  Severe AEs | 0 | 0
  Moderate AEs | 1 | 0
  Mild AEs | 12 | 8

4. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight after 6 weeks of treatment
Time Frame: Week 0, Week 6
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. Missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
kg | 0.09 (0.79) | -0.10 (0.99)

5. Secondary Outcome: Electrocardiogram (ECG) Worsening
Description: The number of subjects having an electrocardiogram (ECG) that changed from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant'. 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Week 0, Week 6
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
participants | 2 | 0

6. Secondary Outcome: Diastolic BP (Blood Pressure)
Description: Values at baseline (Week 0) and at Week 6
Time Frame: Week 0, Week 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
mmHg
  Week 0 (Baseline) | 77.3 (11.1) | 75.4 (11.1)
  Week 6 | 76.8 (10.4) | 76.7 (10.0)

7. Secondary Outcome: Systolic BP (Blood Pressure)
Description: Values at baseline (Week 0) and at Week 6
Time Frame: Week 0, Week 6.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIAC | Mix30
Number analyzed (Participants) | 33 | 32
mmHg
  Week 0 (Baseline) | 137.5 (15.5) | 130.8 (17.4)
  Week 6 | 137.0 (17.0) | 130.9 (16.0)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 6 weeks + 5 days follow up.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | SIAC | Mix30
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/32
Other Adverse Events (participants affected / at risk) | 5/33 | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIAC (N=33) | Mix30 (N=32)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIAC (N=33) | Mix30 (N=32)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.